CLINICAL TRIAL: NCT01382927
Title: Impact of Spontaneous Breathing on Ventilation Distribution in Obese Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Oliver C. Radke, MD, PhD, DEAA, Dpt of Anesthesia and Perioperative Care
Other Study IDs: SBVOBP
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Obesity; Hip Arthroplasty; General Anesthesia; Spinal Anesthesia; Atelectasis
MeSH Terms: conditions — Obesity; Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- General Anesthesia
- Spinal Anesthesia

SUMMARY:
General anesthesia (GA) and paralysis are factors which facilitate atelectasis formation, especially in obese patients. Spontaneous breathing can reduce the amount of atelectasis. In this study, the investigators are comaparing obese patients undergoing hip arthroplasty in GA versus spinal anesthesia. Distribution of ventilation during and after anesthesia is assessed by eletrical impedance tomography (EIT).

ELIGIBILITY:
Inclusion Criteria:

* BMI >30
* age 18-85
* elective hip arthroplasty in general anesthesia or spinal anesthesia

Exclusion Criteria:

* pregnancy/breastfeeding
* allergies against drugs used for the anesthesia
* contraindications for EIT
* severe cardiac or pulmonary comorbidities
* unable to consent or understand/follow study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese Patients aged 18-85, scheduled for elective hip arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2011-04

PRIMARY OUTCOMES:
arterial pO2 on room air | 24hrs
Center of Ventilation | 24hrs
  measured by EIT

SECONDARY OUTCOMES:
Peak Flow | 24hrs

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Carl-Gustav-Carus, Dresden, Germany, Germany